CLINICAL TRIAL: NCT07187804
Title: Long Term Efficacy of Faricimab Using a Treat and Extend Regimen for Type 3 Macular Neovascularization
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kim's Eye Hospital (Other)
Responsible Party: Principal Investigator, Jae Hui Kim, Director of Clinical Research, Kim's Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-07-004
Record Dates: First submitted 2025-09-13; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Age-related Macular Degeneration (ARMD); Choroidal Neovascularization; Anti-vascular Endothelial Growth Factor
Keywords: Age-related macular degeneration; Type 3 macular neovascularization; Retinal angiomatous proliferation; Faricimab; Treat and extend
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Faricimab treatment arm (Experimental)
  Interventions: Drug: Intravitreal faricimab injection

INTERVENTIONS:
Drug: Intravitreal faricimab injection — * Initial loading injections : every 4 weeks by 12weeks
  * Treat and extend injection(~76 week) : Week 20 - Week 76
  TAE is initiated with a minimum injection interval of 8 weeks. If no recurrence is observed, the interval is extended by 2 weeks at a time, up to a maximum of 16 weeks. In the event of recurrence, the injection interval is reduced to 8 weeks, regardless of the previous schedule. The minimum injection interval remains 8 weeks.

SUMMARY:
Type 3 macular neovascularization (MNV) is a subtype of neovascular age-related macular degeneration accounting for 10-20% of cases, notable for high rates of bilateral involvement and risk of profound vision loss, particularly if undertreated. Early and proactive therapy is crucial to prevent progression and preserve vision.

Faricimab offers potential advantages in this setting. Eyes with type 3 MNV often show thin choroid, reticular pseudodrusen, and high GA risk, reflecting compromised choroidal perfusion. While anti-vascular endothelial growth factor (VEGF) agents suppress neovascularization, prolonged VEGF blockade may impair choriocapillaris health. Ang-2 inhibition, by promoting Tie2 activation and vascular stability, may protect choriocapillaris and reduce widespread retinal edema and hemorrhages observed in type 3 MNV.

Finally, while treat-and-extend is widely used in practice, existing trials (TENAYA, LUCERNE) applied broader extension intervals than typically used clinically. In type 3 MNV, where undertreatment carries severe consequences, a more stringent faricimab-based treat-and-extend regimen with 2-week interval adjustments warrants investigation.

DETAILED DESCRIPTION:
1.1 The Nature of Type 3 macular neovascularization (MNV) and Recommended Therapeutic Approaches Type 3 MNV, also known as retinal angiomatous proliferation is a subtype of neovascular age-related macular degeneration (AMD) that is characterized by intraretinal neovascularization. The incidence of type 3 neovascularization is relatively lower than other subtypes of neovascular AMD, constituting 10 to 20% of entire neovascular AMD. However, it is a very important disorder because it often leads bilateral visual deterioration. The high risk of bilateral involvement is characteristic of type 3 neovascularization. In some cases, the visual prognosis of the initially uninvolved eye with better vision, is poorer than the initially involved eye. In addition, profound visual loss may occur during the treatment course, especially in undertreated cases.

Thus, preserving vision is particularly important in type 3 neovascularization, which subsequently highlights the importance of investigating more effective treatment strategies. We previously suggested the need for proactive treatment in type 3 neovascularization to reduce the risk of abrupt visual loss. Furthermore, due to the progressive nature of type 3 MNV, there is an increased risk of visual impairment as the stages advance. Therefore, it is imperative to administer aggressive treatment during the early phase of the disorder to impede the progression of disease stages.

1.2 Why is Faricimab Particularly Advantageous for Type 3 MNV? (My own hypothesis) 1.2.1 The potential of ang-2 inhibition in preserving choriocapillaris Eyes with type 3 MNV usually exhibits very thin choroid, a high prevalence of reticular pseudodrusen, and a lack of choroidal vascular hyperpermeability. These observations collectively indicate compromised choroidal perfusion in such eyes. In fact, the occurrence of geographic atrophy (GA) is particularly elevated in type 3 MNV, and it serves as a significant contributing factor to the progressive deterioration of visual acuity over the long term in this condition. Due to these factors, maintaining adequate choroidal perfusion becomes particularly crucial in the treatment of type 3 MNV.

The choriocapillaris is the most critical tissue for perfusion into the retinal pigment epithelium and retinal outer layers. While anti-vascular endothelial growth factor (VEGF) therapy is highly effective in stabilizing neovascularization, there have been concerns regarding its potential negative impact on the maintenance of retinal pigment epithelium and choriocapillaris by suppressing physiological VEGF, particularly following aflibercept therapy. In 2016, I was the first to propose the possibility that these aspects could pose a concern in the management of patients with type 3 MNV during actual clinical practice.

It has been demonstrated in animal models of choroidal neovascularization that tie2 activation has the potential to induce choriocapillaris regeneration. It is not yet certain whether such phenomena occur in humans. Nonetheless, these research findings can provide support for the hypothesis that tie2 activation through ang-2 inhibition could potentially confer benefits in cases of compromised choroidal perfusion, such as in type 3 MNV.

1.2.2 The importance of promoting vascular stability in the treatment of type 3 MNV In Type 3 MNV, it is well-known that the neovascular lesion itself is often accompanied by extensive and severe retinal edema disproportionate to its size. Additionally, retinal hemorrhages unrelated to the location of the neovascular lesion can frequently occur. Dr. Richard Spaide, from Vitreous Retina Macula Consultants of New York, has proposed that the rapid elevation of VEGF levels leads to the occurrence of such phenomena, including increased vascular permeability and leakage, not only in the neovascular lesion but also in the surrounding retinal vessels. If this hypothesis is valid, it underscores the potential benefit of ang-2 inhibition in the treatment of type 3 MNV, as it suggests that enhancing overall retinal vessel stability, rather than solely focusing on neovascular lesion suppression, could be of substantial advantage.

1.3 Why is an Additional Treat-and-Extend Study Utilizing Faricimab Deemed Necessary? The treat-and-extend regimen is widely acknowledged as a highly effective and efficient treatment approach for type 3 MNV, and it is extensively utilized in industrialized countries. In the TENEYA and LUCERNE clinical trials, conducted to evaluate the introduction of faricimab, personalized treatment intervals (PTIs) were employed for treatment, and starting from the second year, a treatment approach similar to treat-and-extend was implemented.

This approach offers a better reflection of treatment patterns in real-world settings compared to the fixed-dosing regimen utilized in previous clinical trials for the introduction of other anti-VEGF agents. Moreover, as suggested by Khanani et al., it may maximize the benefits of angiopoietin-2 blockade. However, it still differs slightly from the treat-and-extend approach commonly employed in actual clinical practice. Furthermore, in the case of type 3 MNV where undertreatment can have severe detrimental effects on the prognosis, the approach of extending injection intervals by 4 weeks, as utilized in the TENAYA and LUCERNE studies, may not be appropriate. It is deemed necessary to consider a more stringent injection extension approach with intervals of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

[General]

* Signed Informed Consent Form
* Age > 50 years at the time of signing Informed Consent Form
* Participants who are able to comply with the study protocol, in the investigator's judgment
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception (will be defined in details in protocol)

[Ocular]

* BCVA that is equal or higher than 24 Early Treatment Diabetic Retinopathy Study letters on Screening Day/ Day 0.
* Confirmed diagnosis, by the investigator, of symptomatic type 3 neovascularization based on sufficiently clear ocular media and adequate pupillary dilatation allowing acquisition of good quality retinal images for confirmation.
* Treatment naive participants

Exclusion Criteria:

[General]

* Treatment with investigational therapy (device, drug, or traditional medicine with the exception of vitamins and minerals) within 3 months prior to initiation of study treatment on study Day 1
* Any major illness or major surgical procedure within 1 month before screening
* Active cancer within the 12 months prior to study Day 1 except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of < 6 (Grade Group of 1) and a stable prostate-specific antigen for >12 months
* Continuous use of any medications and treatments (which will be indicated in the Prohibited Therapy section in protocol)
* Systemic treatment for suspected or active systemic infection on study Day 1
* Uncontrolled blood pressure, defined as systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg while the participant is at rest on study Day 1
* History of stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to study Day 1
* History of other disease, metabolic dysfunction, physical examination finding, or historical or current clinical laboratory findings giving reasonable suspicion of a condition that contraindicates the use of the investigational drug or that might affect interpretation of the results of the study or renders the participant at high risk for treatment complications in the opinion of the investigator
* History of severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the faricimab injection, study-related procedure preparations (including fluorescein and indocyanine green dyes), dilating drops, or any of the anesthetic and antimicrobial preparations used by a participant during the study
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 28 days after the final dose of faricimab

[Ocular]

* Significant media opacities, including cataract, in the study eye that might interfere with visual acuity, assessment of safety, or fundus photography.
* Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.

Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.

* Any history of uveitis in either eye.
* Presence of definite chorioretional anastomosis
* Subretinal hemorrhage that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye. (If the blood is under the fovea, then the fovea must be surrounded 270 degrees by visible macular neovascularization.)
* Scar or fibrosis, making up > 50% of total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye.
* Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 76 week study period.
* Prior vitrectomy in the study eye
* Any history of macular hole of stage 2 and above in the study eye.
* Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as it's unlikely to interfere with the injection.
* Prior trabeculectomy or other filtration surgery in the study eye.
* Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye.
* Active intraocular inflammation in either eye.
* Active ocular or periocular infection in either eye.
* Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of an yttrium aluminum garnet [YAG] posterior capsulotomy) in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2028-09-22 (Estimated); Study Completion 2028-09-22 (Estimated)

PRIMARY OUTCOMES:
Change in CST (central subfield thickness) | Baseline to week 76
  Change in central retinal thickness, as measured by optical coherence tomography, from baseline to week 76

SECONDARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | Baseline to week 76
  Change in BCVA from baseline to week 76
Choroidal thickness | Baseline to week 76
  Change in choroidal thickness from baseline to week 76
Geographic atrophy (GA) development | Baseline to week 76
  Proportion of eyes experiencing development of GA from baseline to week 76
Fluid resolution | Week 20, 52, and 76
  Proportion of eyes experiencing complete resolution of retinal fluids at week 20, 52, and 76
Presence of neovascularization | Baseline, week 20, 52, and 76
  Proportion of patients with neovascularization at baseline, week 20, 52, and 76
Number of injection | Baseline to week 76
  Total number of injections from baseline to week 76
Maximum injection interval | Baseline to 76 weeks
  Proportion of patients achieved 12 weeks and 16 weeks injection interval
Adverse event | Baseline to week 76
  Proportion of patients experiencing adverse event during study period

CONTACTS AND LOCATIONS:
Locations (1):
- Kim's Eye Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khanani AM, Guymer RH, Basu K, Boston H, Heier JS, Korobelnik JF, Kotecha A, Lin H, Silverman D, Swaminathan B, Willis JR, Yoon YH, Quezada-Ruiz C. TENAYA and LUCERNE: Rationale and Design for the Phase 3 Clinical Trials of Faricimab for Neovascular Age-Related Macular Degeneration. Ophthalmol Sci. 2021 Nov 17;1(4):100076. doi: 10.1016/j.xops.2021.100076. eCollection 2021 Dec. PMID 36246941
- [Result] Spaide RF. NEW PROPOSAL FOR THE PATHOPHYSIOLOGY OF TYPE 3 NEOVASCULARIZATION AS BASED ON MULTIMODAL IMAGING FINDINGS. Retina. 2019 Aug;39(8):1451-1464. doi: 10.1097/IAE.0000000000002412. PMID 30550528
- [Result] Kim JH, Kim JR, Kang SW, Kim SJ, Ha HS. Thinner choroid and greater drusen extent in retinal angiomatous proliferation than in typical exudative age-related macular degeneration. Am J Ophthalmol. 2013 Apr;155(4):743-9, 749.e1-2. doi: 10.1016/j.ajo.2012.11.001. Epub 2013 Jan 11. PMID 23317655
- [Result] Heier JS, Khanani AM, Quezada Ruiz C, Basu K, Ferrone PJ, Brittain C, Figueroa MS, Lin H, Holz FG, Patel V, Lai TYY, Silverman D, Regillo C, Swaminathan B, Viola F, Cheung CMG, Wong TY; TENAYA and LUCERNE Investigators. Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE): two randomised, double-masked, phase 3, non-inferiority trials. Lancet. 2022 Feb 19;399(10326):729-740. doi: 10.1016/S0140-6736(22)00010-1. Epub 2022 Jan 24. PMID 35085502
- [Result] Kim JH, Kim JW, Kim CG, Lee DW. LONG-TERM CHANGES IN CHOROIDAL THICKNESS IN EYES WITH TYPE 3 MACULAR NEOVASCULARIZATION. Retina. 2021 Jun 1;41(6):1251-1258. doi: 10.1097/IAE.0000000000003010. PMID 33136977
- [Result] Su D, Lin S, Phasukkijwatana N, Chen X, Tan A, Freund KB, Sarraf D. AN UPDATED STAGING SYSTEM OF TYPE 3 NEOVASCULARIZATION USING SPECTRAL DOMAIN OPTICAL COHERENCE TOMOGRAPHY. Retina. 2016 Dec;36 Suppl 1:S40-S49. doi: 10.1097/IAE.0000000000001268. PMID 28005662
- [Result] Kim JH, Kim JW, Kim CG. INCIDENCE AND TIMING OF PIGMENT EPITHELIAL DETACHMENT AND SUBRETINAL FLUID DEVELOPMENT IN TYPE 3 MACULAR NEOVASCULARIZATION ASSOCIATED WITH AGE-RELATED MACULAR DEGENERATION. Retina. 2023 Aug 1;43(8):1264-1273. doi: 10.1097/IAE.0000000000003797. PMID 36977322
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW, Cho SY. DIFFERENCE IN TREATMENT OUTCOMES ACCORDING TO OPTICAL COHERENCE TOMOGRAPHY-BASED STAGES IN TYPE 3 NEOVASCULARIZATION (RETINAL ANGIOMATOUS PROLIFERATION). Retina. 2018 Dec;38(12):2356-2362. doi: 10.1097/IAE.0000000000001876. PMID 29019795
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Prechoroidal Cleft in Type 3 Neovascularization: Incidence, Timing, and Its Association with Visual Outcome. J Ophthalmol. 2018 Nov 19;2018:2578349. doi: 10.1155/2018/2578349. eCollection 2018. PMID 30581602
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Early Recurrent Hemorrhage in Submacular Hemorrhage Secondary to Type 3 Neovascularization or Retinal Angiomatous Proliferation: Incidence and Influence on Visual Prognosis. Semin Ophthalmol. 2018;33(6):820-828. doi: 10.1080/08820538.2018.1511814. Epub 2018 Aug 23. PMID 30136868
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW. Abrupt visual loss during anti-vascular endothelial growth factor treatment for type 3 neovascularization. Int J Ophthalmol. 2019 Mar 18;12(3):480-487. doi: 10.18240/ijo.2019.03.20. eCollection 2019. PMID 30918819
- [Result] Chang YS, Kim JH, Yoo SJ, Lew YJ, Kim J. Fellow-eye neovascularization in unilateral retinal angiomatous proliferation in a Korean population. Acta Ophthalmol. 2016 Feb;94(1):e49-53. doi: 10.1111/aos.12748. Epub 2015 May 17. PMID 25981599
- [Result] Kim JH, Chang YS, Kim JW, Kim CG, Lee DW, Kim HS. LONG-TERM VISUAL CHANGES IN INITIALLY STRONGER FELLOW EYES IN PATIENTS WITH UNILATERAL TYPE 3 NEOVASCULARIZATION. Retina. 2019 Sep;39(9):1672-1681. doi: 10.1097/IAE.0000000000002239. PMID 29979454
- [Result] Yannuzzi LA, Negrao S, Iida T, Carvalho C, Rodriguez-Coleman H, Slakter J, Freund KB, Sorenson J, Orlock D, Borodoker N. Retinal angiomatous proliferation in age-related macular degeneration. Retina. 2001;21(5):416-34. doi: 10.1097/00006982-200110000-00003. PMID 11642370
- [Result] Freund KB, Ho IV, Barbazetto IA, Koizumi H, Laud K, Ferrara D, Matsumoto Y, Sorenson JA, Yannuzzi L. Type 3 neovascularization: the expanded spectrum of retinal angiomatous proliferation. Retina. 2008 Feb;28(2):201-11. doi: 10.1097/IAE.0b013e3181669504. PMID 18301024